CLINICAL TRIAL: NCT06070285
Title: Delving Into the Patterns of Patient Engagement and Trends in Participation Within Recurrent Ovarian Cancer Clinical Trials
Brief Title: Investigating Participation Patterns Among Recurrent Ovarian Cancer Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 72827906
Record Dates: First submitted 2023-09-30; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-09

CONDITIONS: Recurrent Ovarian Cancer
Keywords: Recurrent Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical trials, with a particular focus on recurrent ovarian cancer, play a crucial role in assessing the safety and efficacy of novel treatments for this condition. These trials serve as essential tools to determine whether new medications outperform traditional therapies, providing substantial evidence to support their widespread adoption.

By actively participating in recurrent ovarian cancer observational study serves pivotal role in expanding the boundaries of medical knowledge and advancing the quality of care provided to those enduring the same condition.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old
* Able to comprehend the investigational nature of the protocol and provide informed consent
* Diagnosis of recurrent ovarian cancer

Exclusion Criteria:

* No diagnosis of recurrent ovarian cancer confirmed
* Inability to perform regular electronic reporting
* Patient does not understand, sign, and return consent form

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with recurrent ovarian cancer who are actively considering enrolling in a clinical trial for said condition, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to participate in a recurrent ovarian cancer clinical trial | 3 months
Rate of patients who remain in recurrent ovarian cancer clinical research to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Buechel M, Herzog TJ, Westin SN, Coleman RL, Monk BJ, Moore KN. Treatment of patients with recurrent epithelial ovarian cancer for whom platinum is still an option. Ann Oncol. 2019 May 1;30(5):721-732. doi: 10.1093/annonc/mdz104. PMID 30887020
- [Background] Ozga M, Aghajanian C, Myers-Virtue S, McDonnell G, Jhanwar S, Hichenberg S, Sulimanoff I. A systematic review of ovarian cancer and fear of recurrence. Palliat Support Care. 2015 Dec;13(6):1771-80. doi: 10.1017/S1478951515000127. Epub 2015 Mar 2. PMID 25728373
- [Background] Hilal Z, Schultheis B, Hartmann F, Dogan A, Cetin C, Krentel H, Schiermeier S, Tempfer CB. What Characterizes Long-term Survivors of Recurrent Ovarian Cancer? Case Report and Review of the Literature. Anticancer Res. 2016 Oct;36(10):5365-5371. doi: 10.21873/anticanres.11110. PMID 27798900

DOCUMENTS (1):
  • Informed Consent Form (2023-09-30): https://cdn.clinicaltrials.gov/large-docs/85/NCT06070285/ICF_000.pdf